CLINICAL TRIAL: NCT06633627
Title: Identification and Quantification of Neurological Responses in Patients with Dentine Hypersensitivity
Brief Title: Neurological Responses in Patients with Dentine Hypersensitivity
Status: Recruiting | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other); HALEON (Industry)
Responsible Party: Sponsor
Other Study IDs: STH22405; 230613 (Other Grant/Funding Number: Haleon)
Record Dates: First submitted 2024-10-02; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Dentine Hypersensitivity
Keywords: Electroencephalography; Dentine Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental: Patients with dentine sensitivity
  Interventions: Other: Recording of brain activity using electroencephalography (EEG)
- Control: Patients without dentine sensitivity
  Interventions: Other: Recording of brain activity using electroencephalography (EEG)

INTERVENTIONS:
Other: Recording of brain activity using electroencephalography (EEG) — Electroencephalography (EEG) responses to sensitivity stimuli applied to the teeth in patients with and without dentine hypersensitivity will be compared

SUMMARY:
Dentine hypersensitivity (also known as sensitive teeth) is a common dental condition in which the dentine, a layer of sensitive hard tissue under the enamel of the teeth, becomes exposed making the teeth sensitive to stimuli, such as hot and cold. It poses a significant challenge for clinicians and affects patients' quality of life.

The overall aim of the study is to understand if a way of measuring brain activity (electroencephalography [EEG]) shows a response to tooth stimulation, and see how these responses may be different in patients with dentine sensitivity.

EEG records brain signals and can provide information about how the brain processes painful stimuli. EEG recording is a non-evasive and painless procedure. It involves using a cap with small sensors called electrodes to pick up brain signals. During the EEG assessment appointment, brain signals will be recorded throughout the duration when cold temperatures and short bursts of air are applied to the tooth. Brain signals recorded during tooth stimulation from participants with and without dentine sensitivity will then be compared to explore if there are any differences.

The investigators hope that EEG responses could be helpful to objectively assess dentine sensitivity, further the understanding of brain processing of dental pain, and allow the comparison of the effectiveness of different treatment options in the future.

This information may help to improve treatments and the quality of life for patients with dentine sensitivity and potentially other types of dental pain.

DETAILED DESCRIPTION:
Dentine hypersensitivity (DH) is a common dental condition that has been defined as a 'short, sharp pain arising from exposed dentine in response to stimuli typically thermal, evaporative, tactile, osmotic or chemical and which cannot be ascribed to any other form of dental defect or pathology'. Many DH interventions have been investigated over the last 60 years, but a lack of standardisation of pain measurement and objectivity of measures are major limitations for assessing the efficacy of products (or understanding why products fail). A potential solution to this problem is greater understanding of the pain propagation mechanism from controlled stimulus to objective, measurable markers of pain severity.

EEG (electroencephalography) is a non-invasive technique that measures the electrical activity of the brain using the electrodes placed on the scalp. EEG provides information about the brain's electrical activity over time, helping diagnose and understand certain neurological conditions. The investigators have carried out a number of studies using human dental pulp and other human tissue to further understand the mechanisms of pain including pulpal pain.

Evoked potentials are EEG responses to specific stimuli, such as light, sound or heat. Pain-evoked potentials from tooth pulp are evoked potentials specifically related to pain originating from the pulp of a tooth. This type of measurement records the brain's electrical response to a stimulus applied to a tooth, such as thermal stimuli. The resulting EEG recording can provide information about how the central nervous system processes painful stimuli, including the speed and magnitude of the response. It was hypothesised that EEG pain-evoked potentials, if generated and measured in a controlled and repeatable way, can potentially be used (in conjunction with other diagnostic methods) to objectively evaluate the severity of dentine sensitivity and compare the efficacy of different treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years and older;
2. Understands and is willing, able and likely to comply with all study procedures and restrictions;
3. Accepts the form of the study and signs a declaration of informed consent;
4. In good health (in the opinion of the clinical dental professional);
5. A minimum of 10 teeth not including teeth with crowns or bridges from upper right 4 to upper left 4 and lower right 4 to lower left 4;

For patients with dentine sensitivity only (experimental group): self-reported sensitivity in at least 1 tooth; confirmed by response to air puff.

Exclusion Criteria:

1. Adults currently using maxillary or mandibular orthodontic appliances;
2. Obvious signs of untreated caries, which in the opinion of the clinical dental professional, will affect the scientific validity of the study;
3. Periodontal pocket depth ≥4mm in the anterior upper or lower sextants;
4. Evidence of periodontitis.
5. Have a history of seizures;
6. Taking medications that affect brain responses;
7. Experience damaged skin on the scalp due to cuts, psoriasis, eczema, or other conditions;
8. Any participant who in the investigator's judgment will not comply with the study protocol;
9. Any participant who has difficulties in adequate understanding of English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending routine restorative appointments at Charles Clifford Dental Hospital in Sheffield will be screened as potential eligible participants for the study by members of the direct clinical care team and informed about the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-11 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography (EEG) responses to tooth stimulation | 1 hour
  EEG responses to tooth stimulation will be measured, and EEG responses will be compared between participants with and without sensitive teeth

SECONDARY OUTCOMES:
Correlation between Dentine hypersensitivity experience questionnaire (DHEQ) score and EEG responses | 30 minutes
  Participants will be asked to complete the Dentine Hypersensitivity Experience Questionnaire (DHEQ). The DHEQ has 48 questions of which 34 comprise an impact scale. The DHEQ score is calculated as the sum of the scores from the questions, with a possible range of 34-238. A higher DHEQ score indicates that dentine hypersensitivity has a greater impact on the participant's quality of life.
  DHEQ score will be correlated with EEG responses recorded during tooth stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Boissonade, BDS, PhD, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The summary protocol and results summary will be shared. No identifiable information from the participants will be shared.

REFERENCES:
- [Background] Rodd HD, Boissonade FM. Substance P expression in human tooth pulp in relation to caries and pain experience. Eur J Oral Sci. 2000 Dec;108(6):467-74. doi: 10.1034/j.1600-0722.2000.00924.x. PMID 11153921
- [Background] Rodd HD, Boissonade FM. Innervation of human tooth pulp in relation to caries and dentition type. J Dent Res. 2001 Jan;80(1):389-93. doi: 10.1177/00220345010800011601. PMID 11269734
- [Background] Rodd HD, Boissonade FM. Comparative immunohistochemical analysis of the peptidergic innervation of human primary and permanent tooth pulp. Arch Oral Biol. 2002 May;47(5):375-85. doi: 10.1016/s0003-9969(02)00012-2. PMID 12015218
- [Background] Rodd HD, Boissonade FM. Immunocytochemical investigation of immune cells within human primary and permanent tooth pulp. Int J Paediatr Dent. 2006 Jan;16(1):2-9. doi: 10.1111/j.1365-263X.2006.00682.x. PMID 16364087
- [Background] Biggs JE, Yates JM, Loescher AR, Clayton NM, Boissonade FM, Robinson PP. Vanilloid receptor 1 (TRPV1) expression in lingual nerve neuromas from patients with or without symptoms of burning pain. Brain Res. 2007 Jan 5;1127(1):59-65. doi: 10.1016/j.brainres.2006.10.014. Epub 2006 Nov 14. PMID 17109831
- [Background] Bird EV, Robinson PP, Boissonade FM. Na(v)1.7 sodium channel expression in human lingual nerve neuromas. Arch Oral Biol. 2007 May;52(5):494-502. doi: 10.1016/j.archoralbio.2006.11.011. Epub 2007 Jan 8. PMID 17210118
- [Background] Rodd HD, Boissonade FM, Day PF. Pulpal status of hypomineralized permanent molars. Pediatr Dent. 2007 Nov-Dec;29(6):514-20. PMID 18254423
- [Background] Morgan CR, Bird EV, Robinson PP, Boissonade FM. TRPA1 expression in human lingual nerve neuromas in patients with and without symptoms of dysaesthesia. Neurosci Lett. 2009 Nov 13;465(2):189-93. doi: 10.1016/j.neulet.2009.08.055. Epub 2009 Aug 26. PMID 19715741
- [Background] Kaewpitak A, Bauer CS, Seward EP, Boissonade FM, Douglas CWI. Porphyromonas gingivalis lipopolysaccharide rapidly activates trigeminal sensory neurons and may contribute to pulpal pain. Int Endod J. 2020 Jun;53(6):846-858. doi: 10.1111/iej.13282. Epub 2020 Mar 23. PMID 32058593
- [Background] Solis-Castro OO, Wong N, Boissonade FM. Chemokines and Pain in the Trigeminal System. Front Pain Res (Lausanne). 2021 Jul 9;2:689314. doi: 10.3389/fpain.2021.689314. eCollection 2021. PMID 35295531
- [Background] Azab AM, Ahmadi H, Mihaylova L, Arvaneh M. Dynamic time warping-based transfer learning for improving common spatial patterns in brain-computer interface. J Neural Eng. 2020 Feb 18;17(1):016061. doi: 10.1088/1741-2552/ab64a0. PMID 31860902
- [Background] Arvaneh M, Robertson IH, Ward TE. A P300-Based Brain-Computer Interface for Improving Attention. Front Hum Neurosci. 2019 Jan 4;12:524. doi: 10.3389/fnhum.2018.00524. eCollection 2018. PMID 30662400
- [Background] Hu X, Racek AJ, Bellile E, Nascimento TD, Bender MC, Toback RL, Burnett D, Khatib L, McMahan R, Kovelman I, Ellwood RP, DaSilva AF. Brain Functional Changes before, during, and after Clinical Pain. J Dent Res. 2018 May;97(5):523-529. doi: 10.1177/0022034517750136. Epub 2018 Jan 11. PMID 29324076
- [Background] Schiff T, Dotson M, Cohen S, De Vizio W, McCool J, Volpe A. Efficacy of a dentifrice containing potassium nitrate, soluble pyrophosphate, PVM/MA copolymer, and sodium fluoride on dentinal hypersensitivity: a twelve-week clinical study. J Clin Dent. 1994;5 Spec No:87-92. PMID 8534380
- [Background] Addy, M., Dentine hypersensitivity: new perspectives on an old problem. International Dental Journal, 2002. 52(5): p. 367-375.